CLINICAL TRIAL: NCT03610230
Title: A Randomized Open-label Trial Cross-over Trial of Iron Isomaltoside 1000 (Monofer®) Compared With Iron Sucrose (Venofer®) in Peritoneal Dialysis Patients
Brief Title: Iron Isomaltoside Compared With Iron Sucrosein Peritoneal Dialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult patient recruitment due to COVID-19 epidemic
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Mok Ming Yee, Honary Clinical Assitant Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.7
Record Dates: First submitted 2018-05-31; First posted 2018-08-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Iron Deficiency Anemia Treatment
MeSH Terms: interventions — iron isomaltoside 1000; Ferric Oxide, Saccharated

STUDY DESIGN:
Intervention Model Description: prospective randomized cross-over open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monofer (Experimental): Iron Isomaltoside as a single intravenous dose 1000mg over 60 minutes
  Interventions: Drug: Iron Isomaltoside; Drug: Iron sucrose
- Venofer (Active Comparator): Iron Sucrose 200mg weekly intravenous infusions over 2 hours for 5 weeks
  Interventions: Drug: Iron Isomaltoside; Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron Isomaltoside — Iron Isomaltoside 1000 (Monofer®) consists of iron with a tighter binding to its carbohydrate moiety with less free iron
  Other Names: Monofer
Drug: Iron sucrose — the currently most widely used intravenous iron preparation with good safety profile
  Other Names: Monofer

SUMMARY:
1. To compare patient-reported satisfaction, efficacy and short-term safety profile of Monofer® in a single bolus dose with Venofer® in split doses in the treatment of absolute or functional iron deficiency anemia in patients on PD.
2. To compare patient symptomatology on fatigue after treatment of Monofer® compared with Venofer® .

DETAILED DESCRIPTION:
Anemia is commonly present in patients with end-stage renal failure (ESRF) due to insufficient endogenous erythropoietin production, absolute and functional iron deficiency. With the introduction of recombinant human erythropoietin (rHuEPO) and the accessibility of rHuEPO to dialysis patients in the Hospital Authority Drug Formulary, blood transfusion requirement for the treatment of renal related anemia has been much reduced. However, iron store must also be adequately maintained for effective erythropoiesis. The latest KDIGO guideline for anemia in chronic kidney disease recommends iron therapy either in oral or intravenous form if TSAT is ≤30% and ferritin is ≤500µg/L. Oral iron supplement is the most convenient, but it is less effective compared to intravenous forms, especially in the treatment of functional iron deficiency, and has unfavorable patient tolerability and gastro-intestinal side-effect profiles. Iron sucrose (Venofer®) is the most widely used intravenous iron preparation with good safety profile. An initial course of intravenous iron (e.g. Venofer® 200mg weekly for 5 weeks) is commonly given to iron-deplete patients before consideration of maintenance iron therapy. The absence of a vascular access and the need to return to hospital facilities for regular intravenous infusions made intravenous forms less preferred by patients on peritoneal dialysis (PD). Isomaltoside 1000 (Monofer®) consists of iron with a tighter binding to its carbohydrate moiety with less free iron to cause immunologic reactions, and thus allowing for a larger single-dose administration. This may facilitate better acceptance of intravenous iron by patients on PD. The current literature on the efficacy and safety profile of Monofer® in the treatment of renal-related anemia focus mainly on patients on hemodialysis and patients with non-dialysis dependent chronic kidney disease. There is also a lack of information on patient-reported satisfaction on the use of Monofer®. The objective of the current study is to investigate patient-reported satisfaction, efficacy and short-term safety profile of a single bolus of Monofer® compared to Venofer® in the treatment of both absolute and functional iron deficiency anemia in patients on PD. In the second part of the study, patients with recurrent iron deficiency will be crossed-over to receive treatment of the alternative arm. Similar to the first part of the study, patient-reported satisfaction and treatment efficacy will be compared following the same study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin (Hb) level between 8-12g/dL for the previous 4 weeks prior to screening
* TSAT ≤30% and ferritin ≤500µg/L
* Receiving a stable dose of rHuEPO therapy for the previous 4 weeks prior to screening
* Not on intravenous iron therapy for the previous 4 weeks prior to screening
* Minimum weekly total Kt/V of 1.7
* Able to give informed consent

Exclusion Criteria:

* No evidence of active blood loss or hemolysis
* Untreated Vitamin B12 or folate deficiency
* History of multiple allergies
* Iron overload
* Active acute or chronic infections
* Blood transfusion within the previous 12 weeks
* Uncontrolled malignancy
* Severe hyperparathyroidism (PTH >90 pmol/L)
* Thalassemia or hematological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported treatment satisfaction with Monofer® versus Venofer® | 12 weeks
  Patient-reported satisfaction is measured using three questions assessing the view of patients on the medication treatment on the 3 aspects namely effectiveness, convenience and side-effects on a 5-point Likert scale (5 is the maximum score while 1 is the minimum score) and a question on the overall satisfaction of patients with the medication treatment on a numeric rating scale (0 score indicate extremely dissatisfied up to 10, which indicates extremely satisfied). The 4 subscores will be analysed individually.

SECONDARY OUTCOMES:
Hemoglobin level | 12 weeks
  Hemoglobin level
iron profile | 12 weeks
  Serum iron, ferritin, total iron binding capacity, transferrin saturation
average weekly dose of rHuEPO | 12 weeks
  average weekly dose of rHuEPO
patients' subjective assessment of fatigue | 12 weeks
  Visual Analogue Fatigue Scale - where patients indicate on a horizontal line measuring 100mm (where 0 mm indicates no fatigue and 100 mm point indicates very severe fagitue). The length of the patient's mark from 0mm is measured and is taken as the fatigue score
health-related quality of life | 12 weeks
  Kidney Disease Quality of Life Short Form Version 1.3. It consists of 36 questions addressing quality of life. Scores of these 36 questions are calculated according to the author's manual and subsequently analysed as one final total score. The higher the score, the better the quality of life.
the incidence of treatment-related adverse events of Monofer | 12 weeks
  the number of participants with treatment-related adverse events
patients' subjective assessment of fatigue | 12 weeks
  SF-36 Vitality Scale. Patients were asked in the you during the past 4 weeks how the amount of energy they feel by using 4 questions on the frequency of such feelings a 6-point scale (1 indicates all of the time up to 6 which indicates none of the time). The total score of the 4 questions are averaged for analysis with the lowest score indicating more severe fatigue and the highest score indicating the least fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Ming Yee Mok, MBBS FHKAM, Principal Investigator — The University of Hong Kong
Locations (1):
- Tung Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Participant data is kept confidential and is only open to investigators and co-investigators of the study